CLINICAL TRIAL: NCT04736901
Title: Effect of Prophylactic and Therapeutic Anticoagulants in Egyptian Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Neven Sarhan, Lecturer at Faculty of Pharmacy, Misr International University
Other Study IDs: COVID-Anticoagulants
Record Dates: First submitted 2021-02-01; First posted 2021-02-03 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Covid19; Corona Virus Infection; Hypercoagulability
Keywords: COVID-19; Hypercoagulability; Anticoagulants
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Thrombophilia | interventions — Enoxaparin; Rivaroxaban; apixaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Group 1: Enoxaparin therapeutic dose
  Interventions: Drug: Enoxaparin
- Group 2: Enoxaparin prophylactic dose
  Interventions: Drug: Enoxaparin
- Group 3: Rivaroxaban therapeutic dose
  Interventions: Drug: Rivaroxaban
- Group 4: Rivaroxaban prophylactic dose
  Interventions: Drug: Rivaroxaban
- Group 5: Apixaban therapeutic dose
  Interventions: Drug: Apixaban
- Group 6: Apixaban prophylactic dose
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Enoxaparin — 0.5 mg/kg every 12 hours
  Groups: Group 2
Drug: Enoxaparin — 40 mg/day
  Groups: Group 1
Drug: Rivaroxaban — 10 mg once daily
  Groups: Group 4
Drug: Rivaroxaban — 20 mg once daily
  Groups: Group 3
Drug: Apixaban — 2.5 mg twice daily
  Groups: Group 6
Drug: Apixaban — 5 mg twice daily
  Groups: Group 5

SUMMARY:
Since the end of 2019, Egypt and the whole world have been suffering from the Coronavirus Disease 2019 (COVID-19) pandemic, which is caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). According to the World Health Organization (WHO), since the emergence of this new pandemic, there have been more than 97 million confirmed cases of COVID-19 patients and two million death globally; around 160 thousand of these cases are in Egypt.

Recent clinical investigations found a high incidence of thrombotic complications in these patients, even with the standard anticoagulant thromboprophylaxis.Coronavirus disease 2019 (COVID-19) causes a hypercoagulable state. Among the pathological sequel of COVID-19 infection, is the presence of a micro-thrombi in the pulmonary circulation which was shown in several autopsy studies. This thrombosis is believed to contribute to gas exchange impairment among patients with COVID-19 infection.

Some observational studies have shown anticoagulation benefits with reduced mortality, mainly in patients requiring mechanical ventilation. However, these findings remain uncertain and need to be validated in further studies.

This study is performed to evaluate whether therapeutic anticoagulation could improve COVID-19 patients' clinical outcomes compared to prophylactic anticoagulation in terms of improving gas exchange, reducing the need to maintain mechanical ventilation, shortening hospital admission period and mortality rate as well as recovering D-dimmer levels to its normal values.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years..
2. COVID-19 hospitalized patients with pneumonia proved by chest X-ray or CT scan.
3. Confirmed infection with COVID-19 virus using RT-PCR or strongly suspected to be infected with pending confirmation studies.
4. Prothrombin time/international normalized ratio (INR)<1.5; activated partial thromboplastin time (aPTT)/ratio<1.5, and platelet count greater than 100,000/mm3.

Exclusion Criteria:

1. Age greater than 85 years-old
2. Creatinine clearance (CrCl)<10ml/min.
3. Severe circulatory shock with a dose of norepinephrine higher than 1.0 μg/kg/min.
4. Pregnant women.
5. Recent major surgery or severe trauma in the last 3 weeks or recent hemorrhagic stroke in the last 3 months.
6. Active bleeding, blood dyscrasia such as hemophilia and Von Willebrand factor deficiency.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The current research is including moderate and severe SARS-COV-2 patients receiving the same background treatment for 5 days, following an Institutional protocol for standard of care: hydroxychloroquine 400 mg daily, lopinavir/ritonavir 400/100 mg twice daily or/and remdisivir 200 mg LD then 100 once daily as a maintenance dose and anti-coagulation prophylaxis with enoxaparin subcutaneously once a day if D-dimmer between 500-1000 or enoxaparin therapeutic subcutaneously twice daily if D-dimmer >1000.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in clotting factors level | Two weeks
  Difference in clotting factors levels between baseline during inclusion in the study and before discharge.
Change in gas exchange over time | Two weeks
  Difference between ratio of partial pressure of arterial oxygen (PaO2) to the fraction of inspired oxygen (FiO2) at baseline, and before discharge.
Time to increase in oxygenation | Two weeks
  Time to increase in SpO2/FiO2 of 50 or greater compared to the baseline SpO2/FiO2
Duration of hospitalization | Two weeks
  Length of hospital stay

SECONDARY OUTCOMES:
Monitoring of adverse events | Two weeks
  Any signs or symptoms of bleeding will be monitored daily
In hospital mortality rate | Two weeks
  Death occurrence during hospitalization
Monitoring of hemoglobin levels. | Two weeks
  Difference in hemoglobin levels between baseline during inclusion in the study and before discharge.
Monitoring of platelets levels | Two weeks
  Difference in platelets levels between baseline during inclusion in the study and before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Neven Sarhan, PhD, Principal Investigator — Misr International University
Locations (1):
- Teachers Hospital, Cairo, Please Select, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208